CLINICAL TRIAL: NCT04988061
Title: Result of Proactive Parental Educating and Counselling Towards Follow-ups in Parents Whose Infant Fail Newborn Hearing Screening
Brief Title: Proactive Counselling Towards Follow-ups in Newborn Hearing Screening
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no subjects enrolled
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Pittayapon Pitathawatchai, Assistant professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 64-220-13-1
Record Dates: First submitted 2021-07-28; First posted 2021-08-03 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Hearing Loss; Newborn Morbidity
MeSH Terms: conditions — Hearing Loss | interventions — Counseling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counselling arm (Experimental): Educating and Counselling are provided by a physician. Also, the information about hearing screening results and an appointment date are provided by a physician.
  Interventions: Other: counselling
- standard arm (No Intervention): The information about hearing screening results and an appointment date are provided as a routine by either nurses or nurse assistances who perform the screening test.

INTERVENTIONS:
Other: counselling — Educating and Counselling with personal communication for 10-15 minutes and written information about the importance of early identification and intervention for hearing loss are provided by a physician. Also, the information about hearing screening results and an appointment date are provided by a physician.
  Arms: Counselling arm

SUMMARY:
The study aims to investigate if proactive parental educating and counselling can minimize loss to follow-ups of parents whose infant fail newborn hearing screening.

ELIGIBILITY:
Inclusion Criteria:

* The parents whose infants do not pass hearing screening

Exclusion Criteria:

* The parents whose infants have illnesses and are not ready for hearing screening
* The parents who decide to migrate to other areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with loss to follow-ups in all participants whose infants require follow-ups | 6 months
  A loss to follow-up rate which is calculated from number of participants with loss to follow-ups divided by number of all participants whose infants require follow-ups

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No